CLINICAL TRIAL: NCT00398268
Title: Treatment of Unstable Dislocated Both-Bone Distal Forearm Fractures in Children: A Follow-up Study
Brief Title: Dislocated Unstable Distal Both-Bone Forearm Fractures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colaris, Joost, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: colaris06
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Fracture; Forearm; Distal; Child; Treatment
Keywords: Fracture; Forearm; Distal; Child; Treatment
MeSH Terms: conditions — Fractures, Bone

INTERVENTIONS:
Procedure: Kirschner-wire fixation

SUMMARY:
We create a follow-up study of Kirschner wire fixation of a unstable dislocated distal both-bone forearm fracture.

DETAILED DESCRIPTION:
children who arrive at the emergency unit with a dislocated both-bone distal forearm fracture will be asked to join the trial.

After an unstable reposition, the fracture will be fixated with 2 Kirschner-wires. The arm will be immobilised in above elbow cast during 4 weeks. Outpatient clinic visits till a follow-up of 6 months. During these visits we will investigate: consolidation and dislocation on X-ray, function of both arms, complains in daily living and complications.

ELIGIBILITY:
Inclusion Criteria:

* both-bone forearm fracture
* distal
* dislocated
* unstable after reposition
* age < 16 years

Exclusion Criteria:

* fracture older than 1 week
* no informed consent
* refracture
* open fracture (Gustillo 2 and 3)
* both fractures of type torus

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2006-01

PRIMARY OUTCOMES:
pronation and supination

SECONDARY OUTCOMES:
complications, function, esthetics, complains in daily living, X-rays

CONTACTS AND LOCATIONS:
Overall Officials: joost w colaris, drs, Principal Investigator
Locations (1):
- HAGA, location Juliana Children's Hospital, The Hague, South Holland, Netherlands